CLINICAL TRIAL: NCT06521489
Title: Study of Asymmetrical High Flow Nasal Cannula Oxygenation (HFNCO) vs Standard HFNCO on Cardiac Surgical Patients Postoperatively
Brief Title: Asymmetrical HFNCO vs Standard HFNCO Post Cardiac Surgery Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Stavros Theologou, Principal Investigator, Stavros Theologou, RN, Deputy Nurse in Charge - Cardiac Surgery ICU, MSc, MHM, PhD, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NKUAthensGreece
Record Dates: First submitted 2024-07-11; First posted 2024-07-26 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Group 1, Asymmetrical HFNCO (Active Comparator): The intervention involves implementing the Asymmetrical High Flow Oxygenation Nasal Cannula as an oxygen treatment at Study Group 1. In contrast, oxygen supply was provided via conventional High Flow Nasal Cannula as a standard oxygen patients' treatment
  The first Study Group will include patients on Asymmetrical High Flow Nasal Cannula Oxygenation with initial settings of FiO2=60% and gas flow=60L/min.
  Interventions: Device: Asymmetrical High Flow Nasal Cannula Oxygenation
- Study Group 2, Conventional HFNCO (Active Comparator): The intervention involves implementing High Flow Nasal Cannula Oxygenation as an oxygen treatment in Study Group 2.
  The second Study Group will include patients on Conventional High Flow Nasal Cannula Oxygenation with initial settings of FiO2=60% and gas flow=60L/min.
  Interventions: Device: Conventional High Flow Nasal Cannula Oxygenation
- Control Group (No Intervention): No Intervention: Control group In the third group (control group) all patients will receive oxygen treatment according to the standard practice of our cardiac ICU department, i.e., Venturi mask with FiO2=60% and flow of 12L/min.
  In this group, all patients will receive the usual standard of care, with no other interventions included

INTERVENTIONS:
Device: Asymmetrical High Flow Nasal Cannula Oxygenation — Asymmetrical High Flow Nasal Cannula Oxygenation will be implemented in this study group. (1st study group, 60l/min airflow, 60% fiO2)
  Arms: Study Group 1, Asymmetrical HFNCO
Device: Conventional High Flow Nasal Cannula Oxygenation — Conventional High Flow Nasal Cannula Oxygenation will be implemented in this study group. (2nd study group, 60l/min airflow, 60% fiO2)
  Arms: Study Group 2, Conventional HFNCO

SUMMARY:
High-flow oxygen therapy has been applied after extubation in cardiac surgery patients with a well-known successful efficacy. The current authors plan to conduct a prospective, randomized, controlled study of the Asymmetrical device Nasal Cannula High Flow Oxygenation (HFNCO) application on high flow (60L/min) with 60% fiO2 administration versus Conventional device Nasal Cannula High Flow Oxygenation (HFNCO) application on high flow (60L/min) with 60% fiO2 administration and versus Conventional oxygen treatment (Venturi mask) after extubation of patients undergoing elective or non-elective cardiac surgery.

DETAILED DESCRIPTION:
Over the last decade, High Flow Nasal Cannula Oxygenation,(HFNCO) has proven successfully its capability in the management of hypoxemic respiratory failure patients post cardiac surgery. Efficient oxygenation has been recorded in meta-analyses on study population research with BMI > 30 . Moreover, in a recent meta-analysis, it has been documented that the use of HFNCO required less need for upgrade of respiratory support . Similar findings were documented in a study of two different variations of HFNCO treatment as compared with Conventional oxygen therapy (Venturi mask) .

A modified version (Asymmetrical) of HFNCO came on the surface recently whereas the (L) nasal prong has a larger diameter compared with the (R) prong of the nasal cannula.

Research results on hypoxemic patients and laboratory models also revealed interesting measurements on specific respiratory parameters such as minute volume ventilation, respiratory rate, and work of breathing as compared with conventional HFNCO. In addition, there were documented higher resistance flow rates which achieved higher PEEP rates in favor of lung alveoli.

On the other hand, there exists documentation with positive aspects that support the use of a non-rebreathing mask / Venturi mask or surgical mask fixed on top of nasal prongs of HFNCO to augment the fiO2 which finally ends up on the patient.

Aim of the study. The primary goal of the study is the efficacy of the Asymmetrical HFNCO on cardiac surgical patients post-extubation as compared with Conventional HFNCO The secondary goal of the study is the comparison of initial Asymmetrical HFNCO parameters versus a) the avoidance of upgrading Asymmetrical HFNCO supported by a non-rebreathing mask fixed on top of that, versus b) the avoidance of upgrading Asymmetrical HFNCO to Non-Invasive Ventilation (NIV).

The tertiary goal of the study is the comparison of all three patient groups; a) Asymmetrical HFNCO, 60L/min, FiO2 60%, b) Conventional HFNCO 60l/min, FiO2 60%, c) Conventional oxygen therapy Venturi mask 12l/min, FiO2 60% regarding the use of treatment on patients with ΒΜΙ > 30 and regarding respiratory parameters (respiratory rate, pO2/ FiO2, spO2, use of accessory muscles, dyspnoea, comfort and tolerance by using the visual analog scale).

Additional goals of the study are to compare all three patient groups regarding ICU Length of Stay, Hospital Length of Stay, rates of ICU re-admission and re-intubation, and any other respiratory / non-respiratory complications and adverse events ( respiratory-chest infection, pneumothorax, delirium, grand mal, acute renal failure, major bleeding - tamponade, cardiac arrest) . Moreover, the rate of failure of the initial treatment will be recorded (as a major measure of treatment efficacy).

Method This is a prospective, non-blinded, randomized study in post-extubated cardiac surgery patients. The study population will consist of three patient groups;

1. Asymmetrical HFNCO, 60l/min, FiO2 60%,
2. Conventional HFNCO 60l/min, FiO2 60%,
3. Conventional oxygen therapy Venturi mask 12l/min, FiO2 60%

Treatment "failure" will be defined as any crossover from one treatment to another due to the patient's respiratory distress and discomfort. To be more specific, switch from Asymmetrical HFNCO to Conventional HFNCO, or switch from Asymmetrical HFNCO to Conventional oxygen therapy supported by a non-rebreathing mask fixed on top of a nasal cannula, or need for more advanced respiratory support such as non-invasive ventilation or invasive mechanical ventilation

Any implemented treatment would also be defined as "failure" when any irreversible (for at least 48 hours) FiO2/gas-mixture flow escalation might be needed, either it is being recorded in study groups 1 & 2 or control group.

"Failure" would also defined as any irreversible (> 48 hours) crossover from either the HFNCO group to standard practice (Venturi mask) or the need for more advanced respiratory support such as non-invasive ventilation or invasive mechanical ventilation.

An initial power analysis was based on a predicted, average failure rate of 15% in the HFNCO groups and a failure rate of 51% in the control group; this analysis yielded the need for enrollment of a total of 41 HFNCO patients and 21 controls for alpha = 0.05 and power=0.80. To ensure equal numbers of patients in each one of the 2 HFNCO groups, the authors decided to enroll 42 HFNCO patients (n=21 for each NHF group) and 21 controls, resulting in a total enrollment of 63 patients

ELIGIBILITY:
Inclusion Criteria:

* Cardiac ICU adult patients
* >18 years
* After elective or urgent cardiac surgery
* Successful Spontaneous Breathing Trial (SBT) with T-piece and FiO2=60%.
* pO2/ FiO2 <150
* Hemodynamically stable (160>SAP>90mmHg)

Exclusion Criteria:

* Obstructive Sleep Apnea Syndrome supported by CPAP mask on ventilator
* COPD, officially diagnosed, respiratory failure - on exacerbation with serum blood pH <7,35.
* Patients with tracheostomy,
* DNR status,
* Glasgow Coma Scale score < 13,
* Insufficient knowledge of the Greek Language
* Visual or hearing impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Successful weaning (i.e. absence of treatment failure) from Asymmetrical Nasal Cannula High Flow Oxygenation post-extubation from cardiac surgery within at least 48 hours | Up to at least 48 hours post extubation or until ICU discharge (predicted cardiothoracic ICU stay could occasionally extend up to 7 days)]
  Successful weaning (i.e. absence of treatment failure as further described in methods) would be defined as = 0 when there would be avoided successfully any alternation with Conventional Nasal Cannula High Flow Oxygenation, Non Invasive Ventilation, or re-intubation
  For all groups: Unsuccessful weaning (i.e. actual treatment failure as further described in methods) would be defined as =1 when there would not be avoided any alternation with Conventional Nasal Cannula High Flow Oxygenation, Non Invasive Ventilation or re-intubation.

SECONDARY OUTCOMES:
Successful maintenance of Respiration rate within the normal range (12-20/min) on initial airflow at 60 L/min, 60% fiO2 on Asymmetrical Nasal Cannula High Flow Oxygenation | Up to at least 48 hours post extubation or until ICU discharge (predicted cardiothoracic ICU stay could occasionally extend up to 7 days)]
  Successful maintenance of Respiratory rate within normal range would be defined as = 0. Unsuccessful (=1) if exceeds normal range (12-20/min).
  Continuous monitoring and recording of implementation of airflow at 60L/min, 60% fiO2 on Asymmetrical Nasal Cannula High Flow Oxygenation
Successful maintenance of Respiration rate within the normal range (12-20/min) on the initial airflow of 60 L/min, 60% fiO2 with Conventional Nasal Cannula High-Flow Oxygenation | Up to at least 48 hours post extubation or until ICU discharge (predicted cardiothoracic ICU stay could occasionally extend up to 7 days)]
  Successful maintenance of Respiratory rate within normal range would be defined as = 0. Unsuccessful (=1) if exceeds normal range (12-20/min).
  Continuous monitoring and recording of implementation of airflow at 60L/min, 60% fiO2 on Conventional Nasal Cannula High Flow Oxygenation
Successful maintenance of Respiration rate within normal range (12-20/min) with Venturi mask , FiO2: 60%, 15L/min | Up to at least 48 hours post extubation or until ICU discharge (predicted cardiothoracic ICU stay could occasionally extend up to 7 days)]
  Successful maintenance of Respiratory rate within normal range would be defined as = 0. Unsuccessful (=1) if exceeds normal range (12-20/min).
  Continuous monitoring and recording of implementation of Venturi mask, FiO2: 60%, 15L/min
Recording of pO2/FiO2 ratio with initial air flow at 60 L/min & 60% fiO2 with Asymmetrical Nasal Cannula High Flow Oxygenation | Up to at least 48 hours post extubation or until ICU discharge (predicted cardiothoracic ICU stay could occasionally extend up to 7 days)]
  Continuous monitoring and recording of implementation of Asymmetrical Nasal Cannula High Flow Oxygenation with airflow at 60 L/min & 60% fiO2
Recording of pO2/FiO2 ratio with initial airflow at 60 L/min & 60% fiO2 with Conventional Nasal Cannula High Flow Oxygenation | Up to at least 48 hours post extubation or until ICU discharge (predicted cardiothoracic ICU stay could occasionally extend up to 7 days)]
  Continuous monitoring and recording of implementation of Conventional Nasal Cannula High Flow Oxygenation with airflow at 60 L/min & 60% fiO2
Recording of pO2/FiO2 ratio with Venturi mask, 60% fiO2, 12l/min | Up to at least 48 hours post extubation or until ICU discharge (predicted cardiothoracic ICU stay could occasionally extend up to 7 days)]
  Continuous monitoring and recording of implementation of Venturi mask, 60% fiO2, 12l/min
Successful maintenance of saturation O2 in Hemoglobulin within normal range with initial airflow at 60 L/min & 60% fiO2 on Asymmetrical Nasal Cannula High Flow Oxygenation | Up to at least 48 hours post extubation or until ICU discharge (predicted cardiothoracic ICU stay could occasionally extend up to 7 days)]
  Successful maintenance of saturation O2 in Hemoglobulin > 92% would be defined as = 0.
  If saturation O2 < 92 %, it would be defined as Unsuccessful = 1. Continuous monitoring and recording of implementation of initial airflow at 60 L/min & 60% fiO2 on Asymmetrical Nasal Cannula High Flow Oxygenation
Successful maintenance of saturation O2 in Hemoglobulin within normal range with initial airflow at 60 L/min & 60% fiO2 on Conventional Nasal Cannula High Flow Oxygenation | Up to at least 48 hours post extubation or until ICU discharge (predicted cardiothoracic ICU stay could occasionally extend up to 7 days)]
  Successful maintenance of saturation O2 in Hemoglobulin > 92% would be defined as = 0.
  If saturation O2 < 92 %, it would be defined as Unsuccessful = 1. Continuous monitoring and recording of implementation of initial airflow at 60 L/min & 60% fiO2 on Conventional Nasal Cannula High Flow Oxygenation
Successful maintenance of saturation O2 in Hemoglobulin within normal range with Venturi mask, 60% fiO2, 12l/min | Up to at least 48 hours post extubation or until ICU discharge (predicted cardiothoracic ICU stay could occasionally extend up to 7 days)]
  Successful maintenance of saturation O2 in Hemoglobulin > 92% would be defined as = 0.
  If saturation O2 < 92 %, it would be defined as Unsuccessful = 1. Continuous monitoring and recording of implementation of Venturi mask, 60% fiO2, 12l/min
Mobilization of accessory respiratory muscles with initial airflow at 60 L/min & 60% fiO2 on Asymmetrical Nasal Cannula High Flow Oxygenation | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Success would be defined as = 0 when there would be no mobilization of accessory respiratory muscles. Failure would be defined as = 1 when there would be recorded any mobilization and use of accessory respiratory muscles.
  Continuous monitoring and recording of implementation of initial airflow at 60 L/min & 60% fiO2 on Asymmetrical Nasal Cannula High Flow Oxygenation
Mobilization of accessory respiratory muscles with initial airflow at 60 L/min & 60% fiO2 on Conventional Nasal Cannula High Flow Oxygenation. | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Success would be defined as = 0 when there would be no mobilization of accessory respiratory muscles. Failure would be defined as = 1 when there would be recorded any mobilization and use of accessory respiratory muscles.
  Continuous monitoring and recording of implementation of initial airflow at 60 L/min & 60% fiO2 on Conventional Nasal Cannula High Flow Oxygenation.
Mobilization of accessory respiratory muscles with Venturi mask, 60% fiO2, 12l/min | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Success would be defined as = 0 when there would be no mobilization of accessory respiratory muscles. Failure would be defined as = 1 when there would be recorded any mobilization and use of accessory respiratory muscles.
  Continuous monitoring and recording of implementation of Venturi mask, 60% fiO2, 12l/min
Comfort and tolerance of treatment with Visual Analogue Scale on Asymmetrical Nasal Cannula High Flow Oxygenation with initial airflow at 60 L/min & 60% fiO2 | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  To monitor and record a patient's comfort with the Visual Analogue Scale diagnostic tool on a scale of 1 to 10. The patients would give the number 10 should they feel comfortable with their respiratory function and have no difficulty breathing. Number 10 on the Scale would mean the best outcome and number 1 would mean the worst outcome respectively
Comfort and tolerance of treatment with Visual Analogue Scale on Conventional Nasal Cannula High Flow Oxygenation with initial airflow at 60 L/min & 60% fiO2 | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  To monitor and record a patient's comfort with the Visual Analog Scale diagnostic tool on a scale of 1 to 10. The patients would give the number 10 should they feel comfortable with their respiratory function and have no difficulty breathing. Number 10 on the Scale would mean the best outcome and number 1 would mean the worst outcome respectively
Comfort and tolerance of treatment with Visual Analogue Scale with Venturi mask, 60% fiO2, 12l/min | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  To monitor and record a patient's comfort with the Visual Analog Scale diagnostic tool on a scale of 1 to 10. The patients would give the number 10 should they feel comfortable with their respiratory function and have no difficulty breathing. Number 10 on the Scale would mean the best outcome and number 1 would mean the worst outcome respectively
Length of Stay in the ICU | Post cardiothoracic ICU admission period up to 48 hours or untiI actual cardiothoracic ICU discharge]
  There will be recorded the total length of stay in the ICU since admission post surgery
Length of Stay in the Hospital | Post cardiothorasic ICU admission period up to actual hospital discharge
  There will be recorded the total length of stay in the hospital since ICU admission
Number of participants with death in the cardiothoracic ICU post extubation | Post cardiothoracic ICU admission period up to 48 hours or untiI actual cardiothoracic ICU discharge]
  There will be recorded the number of participants that will pass away post extubation in the ICU
Number of participants with Atrial Fibrillation in the ICU post extubation | Post cardiothoracic ICU admission period up to 48 hours or untiI actual cardiothoracic ICU discharge]
  There will be recorded the number of participants that will present Atrial Fibrillation post extubation in the ICU
Number of participants with any Adverse Events in the ICU (respiratory-chest infection, pneumothorax, delirium, grand mal, acute renal failure, major bleeding - tamponade ) | Post cardiothoracic ICU admission period up to 48 hours or untiI actual cardiothoracic ICU discharge]
  There will be recorded the number of participants that will present any Adverse Events (respiratory-chest infection, pneumothorax, delirium, grand mal, acute renal failure, tamponade ) post extubation in the ICU
Number of participants with any Adverse Events in the Hospital (respiratory-chest infection, pneumothorax, delirium, grand mal, acute renal failure, major bleeding - tamponade, cardiac arrest ) | Post cardiothorasic ICU admission period up to 3 months or until actual Hospital discharge
  There will be recorded the number of participants that will present any Adverse Events (respiratory-chest infection, pneumothorax, delirium, grand mal, acute renal failure, tamponade, cardiac arrest) in the Hospital
Percentage of participants presenting unsuccessful (failed) implementation of Asymmetrical Nasal Cannula High Flow Oxygenation treatment | Post cardiothoracic ICU admission period up to 48 hours or untiI actual cardiothoracic ICU discharge]
  There will be recorded the number of participants who will fail to comply with the treatment due to failing to maintain their respiratory parameters within normal range, or due to presenting intolerance and discomfort to the implementation of Asymmetrical Nasal Cannula High Flow Oxygenation treatment
Percentage of participants presenting unsuccessful (failed) implementation of Conventional Nasal Cannula High Flow Oxygenation treatment | Post cardiothoracic ICU admission period up to 48 hours or untiI actual cardiothoracic ICU discharge]
  There will be recorded the number of participants who will fail to comply with the treatment due to failing to maintain their respiratory parameters within normal range, or due to presenting intolerance and discomfort to the implementation of Conventional Nasal Cannula High Flow Oxygenation treatment
Percentage of participants presenting unsuccessful (failed) implementation of Venturi mask oxygen therapy | Post cardiothoracic ICU admission period up to 48 hours or untiI actual cardiothoracic ICU discharge]
  There will be recorded the number of participants who will fail to comply with the treatment due to failing to maintain their respiratory parameters within normal range, or due to presenting intolerance and discomfort to the implementation of Venturi mask oxygen therapy
Number of participants with re-intubation in the ICU | Post cardiothorasic ICU admission period up to 3 months or until actual Hospital discharge
  There will be recorded the number of participants that will be re-intubated due to deterioration of their respiratory parameters.

CONTACTS AND LOCATIONS:
Overall Officials: SPYRIDON A. MENTZELOPOULOS, MD, Study Director — Evangelismos General Hospital of Athens
Locations (1):
- Evangelismos General Hospital of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shiho D, Kusaka Y, Nakano S, Umegaki O. The short-term efficacy of high flow nasal oxygen therapy on cardiovascular surgical patients: a randomized crossover trial. BMC Anesthesiol. 2022 Oct 29;22(1):331. doi: 10.1186/s12871-022-01883-3. PMID 36309660
- [Background] Wang Y, Zhu J, Wang X, Liu NA, Yang Q, Luan G, Ma X, Liu J. Comparison of High-flow Nasal Cannula (HFNC) and Conventional Oxygen Therapy in Obese Patients Undergoing Cardiac Surgery: A Systematic Review and Meta-analysis. In Vivo. 2021 Sep-Oct;35(5):2521-2529. doi: 10.21873/invivo.12533. PMID 34410938
- [Background] Zhu Y, Yin H, Zhang R, Wei J. High-flow nasal cannula oxygen therapy vs conventional oxygen therapy in cardiac surgical patients: A meta-analysis. J Crit Care. 2017 Apr;38:123-128. doi: 10.1016/j.jcrc.2016.10.027. Epub 2016 Nov 9. PMID 27886577
- [Background] Boscolo A, Pettenuzzo T, Zarantonello F, Sella N, Pistollato E, De Cassai A, Congedi S, Paiusco I, Bertoldo G, Crociani S, Toma F, Mormando G, Lorenzoni G, Gregori D, Navalesi P. Asymmetrical high-flow nasal cannula performs similarly to standard interface in patients with acute hypoxemic post-extubation respiratory failure: a pilot study. BMC Pulm Med. 2024 Jan 8;24(1):21. doi: 10.1186/s12890-023-02820-x. PMID 38191347
- [Background] Slobod D, Spinelli E, Crotti S, Lissoni A, Galazzi A, Grasselli G, Mauri T. Effects of an asymmetrical high flow nasal cannula interface in hypoxemic patients. Crit Care. 2023 Apr 18;27(1):145. doi: 10.1186/s13054-023-04441-6. PMID 37072854
- [Background] Montiel V, Robert A, Robert A, Nabaoui A, Marie T, Mestre NM, Guillaume M, Laterre PF, Wittebole X. Surgical mask on top of high-flow nasal cannula improves oxygenation in critically ill COVID-19 patients with hypoxemic respiratory failure. Ann Intensive Care. 2020 Sep 29;10(1):125. doi: 10.1186/s13613-020-00744-x. PMID 32990864
- [Background] Egan B, Sharples AP. Molecular responses to acute exercise and their relevance for adaptations in skeletal muscle to exercise training. Physiol Rev. 2023 Jul 1;103(3):2057-2170. doi: 10.1152/physrev.00054.2021. Epub 2022 Nov 17. PMID 36395350
- [Background] Vieira F, Bezerra FS, Coudroy R, Schreiber A, Telias I, Dubo S, Cavalot G, Pereira SM, Piraino T, Brochard LJ. High Flow Nasal Cannula compared to Continuous Positive Airway Pressure: a bench and physiological study. J Appl Physiol (1985). 2022 May 5. doi: 10.1152/japplphysiol.00416.2021. Online ahead of print. PMID 35511720
- [Result] Theologou S, Ischaki E, Zakynthinos SG, Charitos C, Michopanou N, Patsatzis S, Mentzelopoulos SD. High Flow Oxygen Therapy at Two Initial Flow Settings versus Conventional Oxygen Therapy in Cardiac Surgery Patients with Postextubation Hypoxemia: A Single-Center, Unblinded, Randomized, Controlled Trial. J Clin Med. 2021 May 12;10(10):2079. doi: 10.3390/jcm10102079. PMID 34066244